CLINICAL TRIAL: NCT03161678
Title: Impact of Genetic Variation in CES1 on Antiplatelet Therapy
Brief Title: CES1 Crossover Trial of Clopidogrel and Ticagrelor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Joshua Lewis, Associate Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00074967
Record Dates: First submitted 2017-05-18; First posted 2017-05-22 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction; Thrombosis; Platelet Dysfunction
Keywords: Pharmacogenetics; Carboxylesterase 1 (CES1); Antiplatelet therapy
MeSH Terms: conditions — Myocardial Infarction; Thrombosis | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Ninety healthy Amish subjects (30 CES1 G143E allele carriers, 30 carriers of a risk variant to be determined, and 30 age/sex-matched controls) will be enrolled. We will prospectively evaluate the effect of CES1 genotype on clopidogrel and ticagrelor response, as assessed by agonist-stimulated platelet aggregation, through the completion of a randomized crossover study of clopidogrel (75 mg per day for 7 d) and ticagrelor (90 mg twice daily for 7 d) in 90 healthy Amish individuals stratified by CES1 genotype as described above, with at least a 14-day washout period between drug interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Wild-Type Genotype (Active Comparator): Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Carriers of the CES1 G143E Mutation (Experimental): Research subjects who carry the CES1 G143E allele (rs71647871) will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Carriers of CES1 rs7498748 Mutation (Experimental): Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Other Names: Plavix
Drug: Ticagrelor — Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Other Names: Brilinta

SUMMARY:
The purpose of this investigation is to evaluate when genetic variation in the carboxylesterase 1 (CES1) gene influences antiplatelet therapy response, as assessed by ex vivo platelet aggregometry, in healthy participants treated with clopidogrel and ticagrelor. We hypothesize that genetic variation in CES1 will significantly impact on-clopidogrel platelet aggregation while having a minimal effect in ticagrelor-treated subjects.

Specific Aim: To conduct a prospective randomized crossover study of clopidogrel and ticagrelor in healthy individuals stratified by CES1 genotype. Participants will be recruited by CES1 genotype into a randomized crossover study of clopidogrel (75 mg daily for 7d) and ticagrelor (90 mg twice daily for 7d) with extensive phenotyping including ex vivo platelet aggregometry performed pre- and post-drug administration in order to assess the interaction of genotype and drug choice on on-treatment platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Of Amish descent
* Age 18 to 75 years
* Participant in the Phamacogenomics of Anti-Platelet Intervention (PAPI-1) Study or other Amish Research Center study, or a family member of an Amish Research Center study participant.

Exclusion Criteria:

* Clopidogrel or ticagrelor allergy
* Platelet count < 100,000 mm3 or > 500,000 mm3
* Hematocrit (Hct) < 32% or > 50%
* Blood pressure > 160/95 mm Hg
* Co-existing malignancy
* Creatinine > 2.0 mg/dl
* Aspartate transaminase (AST) or alanine transaminase (ALT) > 2 times the upper limit of normal
* Thyroid-stimulating hormone (TSH) < 0.40 or > 5.50 mU/L
* Pregnant or breast feeding
* History of gastrointestinal bleeding, a major life-threatening bleeding event, active pathological bleeding, bleeding diathesis, or coagulopathy
* History of stroke or transient ischemic attack, deep vein thrombosis, or atrial fibrillation
* History of myocardial infarction, coronary artery bypass surgery, unstable angina, or angioplasty
* History of sick sinus syndrome, 2nd or 3rd degree atrioventricular block, or bradycardia-related syncope
* Type 1 or Type 2 diabetes mellitus
* Surgery in the past 3 months or planned surgery in the next 3 months
* Participant cannot willingly and safely discontinue medications that, in the opinion of the study physician would affect the outcomes to be measured for at least 1 week prior to study initiation through completion of the study
* Participant is unwilling to discontinue taking vitamins and/or supplements that, in the opinion of the study physician would affect the outcomes to be measured for 1 week prior to the study initiation through the the completion of the study
* Any other condition that would place prospective participants at unacceptable risk or render them unable to meet the requirements of the protocol in the opinion of the site investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Lewis, PhD, Principal Investigator — University of Maryland
Locations (1):
- Amish Research Clinic, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is possible that deidentified data will be deposited into large public databases as per NIH data sharing policies (e.g. database of Genotypes and Phenotypes [dbGAP], Pharmacogenomics Knowledgebase [PharmGKB]). Data to be shared would include, but not limited to, anthropometric data, study outcome data, and relevant covariate data used in statistical models of association. It is anticipated that data would be available after the completion of the trial. The data will be obtained from the participants and the study-related research procedures.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In our investigation, participants discontinued all vitamins/supplements at least 7 days before their first clinic visit, which is when drug was randomly assigned. Of the 111 enrolled, 11 (3 controls, 1 G143E, and 7 CES1 rs7498748) withdrew prior to clinic visit 1, thus drug was not assigned to those individuals. As such, the number of individuals shown below do not equal 111 (total enrollment number) but instead show the number of individuals who were randomly assigned to a medication (N=100)
Groups:
- Wild-Type Genotype: Clopidogrel First, Then Ticagrelor: Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to receive clopidogrel first followed by ticagrelor
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Wild Type Genotype: Ticagrelor First, Then Clopidogrel: Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to received ticagrelor first followed by clopidogrel
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel First, Then Ticagrelor: Research subjects who carry a CES1 G143E minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to clopidogrel first followed by ticagrelor.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor First, Then Clopidogrel: Research subjects who carry a CES1 G143E minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to ticagrelor first followed by clopidogrel.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel First, Then Ticagrelor: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to clopidogrel first followed by ticagrelor.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor First, Then Clopidogrel: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. This group was randomized to ticagrelor first followed by clopidogrel.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
Period: Intervention 1 (8 Days)
Arm/Group | Wild-Type Genotype: Clopidogrel First, Then Ticagrelor | Wild Type Genotype: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor First, Then Clopidogrel
Started | 17 | 19 | 10 | 12 | 23 | 19
Completed | 16 | 18 | 10 | 9 | 22 | 19
Not Completed | 1 | 1 | 0 | 3 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Period: Washout (14 Days)
Arm/Group | Wild-Type Genotype: Clopidogrel First, Then Ticagrelor | Wild Type Genotype: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor First, Then Clopidogrel
Started | 16 | 18 | 10 | 9 | 22 | 19
Completed | 16 | 18 | 9 | 9 | 20 | 18
Not Completed | 0 | 0 | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2 | 1
Period: Intervention 2 (8 Days)
Arm/Group | Wild-Type Genotype: Clopidogrel First, Then Ticagrelor | Wild Type Genotype: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor First, Then Clopidogrel | Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel First, Then Ticagrelor | Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor First, Then Clopidogrel
Started | 16 | 18 | 9 | 9 | 20 | 18
Completed | 16 | 18 | 9 | 8 | 20 | 18
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants With Wild-Type Genotype: Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- All Participants Who Carried the CES1 G143E Mutation: Research subjects who carry the CES1 G143E allele (rs71647871) will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- All Participants Who Carried the CES1 Functional Mutation: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Total: Total of all reporting groups
Arm/Group | All Participants With Wild-Type Genotype | All Participants Who Carried the CES1 G143E Mutation | All Participants Who Carried the CES1 Functional Mutation | Total
Number analyzed (Participants) | 34 | 17 | 38 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (10.6) | 44.5 (14.2) | 52.1 (12.9) | 49.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 6 | 23 | 45
  Male | 18 | 11 | 15 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 34 | 17 | 38 | 89
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 17 | 38 | 89
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.4 (4.4) | 27.6 (4.7) | 29.0 (4.9) | 28.1 (4.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 118.2 (12.8) | 117.2 (12.0) | 120.2 (13.9) | 118.9 (13.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 73.8 (8.0) | 70.7 (6.8) | 74.0 (7.7) | 73.7 (7.7)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 210.7 (47.0) | 207.9 (56.2) | 208.8 (43.3) | 209.3 (46.8)
Low-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 135.0 (38.4) | 138.7 (49.6) | 132.0 (39.2) | 134.4 (40.7)
High-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 60.4 (18.0) | 52.8 (14.3) | 60.5 (13.3) | 59.0 (15.6)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 61.9 (21.1) | 71.5 (45.4) | 69.4 (41.2) | 66.9 (35.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximal Platelet Aggregation in Response to Clopidogrel
Description: Ex vivo platelet aggregometry was performed in platelet rich plasma (PRP) after stimulation with 20 μM adenosine diphosphate (ADP) at 2 time points (at baseline prior to drug administration and on the 8th day of clopidogrel [75mg/d]). Maximum platelet aggregation is recorded by the platelet aggregometer as a percentage. Data shown below represent the maximum platelet aggregation value obtained at baseline minus the maximum platelet aggregation value obtained after clopidogrel administration. Thus, values recorded below represent changes from baseline at day 8 and the unit is percent maximum aggregation. Higher reported values represent a greater reduction in platelet aggregation while lower reported values signify a smaller reduction in platelet aggregation when comparing baseline and post-clopidogrel visits.
Time Frame: 8 days of exposure to clopidogrel (change from baseline at day 8 reported)
Population: All of the outcome measures in this trial were pre-specified to be analyzed by genotype. Therefore, Arm/Groups are shown by genotype group rather than per medication sequence order. This is consistent with how baseline characteristics are displayed as well.
Measure: Mean (Standard Error); unit: Percent Maximal Platelet Aggregation
Groups:
- Carriers of CES1 Functional Mutation: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
Arm/Group | Wild-Type Genotype | Carriers of the CES1 G143E Mutation | Carriers of CES1 Functional Mutation
Number analyzed (Participants) | 34 | 17 | 38
Percent Maximal Platelet Aggregation | 32.6 (2.7) | 50.8 (2.1) | 35.0 (2.1)
Statistical Analysis 1: Comparison: Wild-Type Genotype vs Carriers of the CES1 G143E Mutation; Change in platelet aggregation was assessed between the wild-type group and the carriers of the CES1 G143E mutation. The null hypothesis is that, following drug intervention, there is no difference in the change in platelet aggregation between genotype groups; Test type: Other — The effect of CES1 genotype on agonist-stimulated change in platelet aggregation was calculated using variance component method that simultaneously adjusted for age, sex, body mass index (BMI), and relatedness among study participants. Relatedness among participants were accounted for by including a polygenic component as a random effect. Please see the Study Protocol and Statistical Analysis Plan document for additional information; p < 0.001, Regression, Linear; All analyses were adjusted for age, sex, body mass index (BMI), and relatedness among study participants
Statistical Analysis 2: Comparison: Wild-Type Genotype vs Carriers of CES1 Functional Mutation; Change in platelet aggregation was assessed between the wild-type group and the carriers of the CES1 functional mutation (rs7498748). The null hypothesis is that, following drug intervention, there is no difference in the change in platelet aggregation between genotype groups; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.24, Regression, Linear; All analyses were adjusted for age, sex, body mass index (BMI), and relatedness among study participants

2. Primary Outcome: Change in Maximal Platelet Aggregation in Response to Ticagrelor
Description: Ex vivo platelet aggregometry was performed in platelet rich plasma (PRP) after stimulation with 20 μM adenosine diphosphate (ADP) at 2 time points (at baseline prior to drug administration and on the 8th day of ticagrelor [90 mg twice daily]). Maximum platelet aggregation is recorded by the platelet aggregometer as a percentage. Data shown below represent the maximum platelet aggregation value obtained at baseline minus the maximum platelet aggregation value obtained after ticagrelor administration. Thus, values recorded below represent changes from baseline at day 8 and the unit is percent maximum aggregation. Higher reported values represent a greater reduction in platelet aggregation while lower reported values signify a smaller reduction in platelet aggregation when comparing baseline and post-ticagrelor visits.
Time Frame: 8 days of independent exposure to ticagrelor (change from baseline at day 8 reported)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent Maximal Platelet Aggregation
Arm/Group | Wild-Type Genotype | Carriers of the CES1 G143E Mutation | Carriers of CES1 Functional Mutation
Number analyzed (Participants) | 34 | 17 | 38
Percent Maximal Platelet Aggregation | 46.1 (1.5) | 47.8 (1.8) | 39.6 (1.9)
Statistical Analysis 1: Comparison: Wild-Type Genotype vs Carriers of the CES1 G143E Mutation; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.75, Regression, Linear; All analyses were adjusted for age, sex, body mass index (BMI), and relatedness among study participants
Statistical Analysis 2: Comparison: Wild-Type Genotype vs Carriers of CES1 Functional Mutation; [analysis description as in outcome 1, analysis 2]; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.011, Regression, Linear; All analyses were adjusted for age, sex, body mass index (BMI), and relatedness among study participants

ADVERSE EVENTS:
Time Frame: During both intervention periods, the washout period, and for 30 days after the final study visit, up to 57 day
Description: Adverse event data were collected during both intervention periods, the washout period, and for 30 days after the final study visit.
Groups:
- Wild-Type Genotype: Clopidogrel: Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who had the wild-type genotype and during the clopidogrel intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Wild Type Genotype: Ticagrelor: Research subjects with wild type CES1 genotypes will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who had the wild-type genotype and during the ticagrelor intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel: Research subjects who carry a CES1 G143E minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who carried the G143E allele and during the clopidogrel intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor: Research subjects who carry a CES1 G143E minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who carried the G143E allele and during the ticagrelor intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who carried the functional mutation (rs7498748) and during the clopidogrel intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
- Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor: Research subjects who carry a CES1 rs7498748 minor allele will be studied before and after oral ingestion of clopidogrel (75 mg/d for 8 days) and ticagrelor (90 mg twice daily for 8 days) treatment. The data shown here are for participants who carried the functional mutation (rs7498748) and during the ticagrelor intervention.
  Clopidogrel: Clopidogrel (75 mg/d for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
  Ticagrelor: Ticagrelor (90 mg twice daily for 8 days) will be administered. Measures of pharmacodynamics will be assessed pre- and post-drug administration.
Arm/Group | Wild-Type Genotype: Clopidogrel | Wild Type Genotype: Ticagrelor | Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel | Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor | Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel | Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/19 | 0/21 | 0/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/19 | 0/21 | 0/41 | 0/39
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 1/19 | 1/21 | 0/41 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wild-Type Genotype: Clopidogrel (N=35) | Wild Type Genotype: Ticagrelor (N=35) | Carboxylesterase 1 (CES1) G143E Mutation: Clopidogrel (N=19) | Carboxylesterase 1 (CES1) G143E Mutation: Ticagrelor (N=21) | Carboxylesterase 1 (CES1) Functional Mutation: Clopidogrel (N=41) | Carboxylesterase 1 (CES1) Functional Mutation: Ticagrelor (N=39)
Knee Pain/Swelling (General disorders) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Knee pain and swelling began after participant started taking clopidogrel 75 mg daily.
Dyspnea (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dyspnea occurred in 1 individual a few days after starting the ticagrelor intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT03161678/Prot_SAP_001.pdf